CLINICAL TRIAL: NCT05377697
Title: The Effect of Lavender Scent Recommended to the Elderly on Sleep Quality and Physical Balance
Brief Title: The Effect of Lavender Scent on Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KaratayUBB
Record Dates: First submitted 2022-04-28; First posted 2022-05-17 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2022-04

CONDITIONS: Sleeping Disorders; Nursing
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry lavender flower scent (Experimental): Participants in the experimental group will be informed about the effects of lavender scent on sleep and lavender sachets will be given. They will be informed that they should put these lavender sachets in their pillows every day and sleep with a lavender sachet for the next month, and that they should not make any changes in their rooms or beds other than the lavender sachet.
  Interventions: Other: Dry lavender flower scent
- Control group (No Intervention): Participants in the control group will not receive any intervention.

INTERVENTIONS:
Other: Dry lavender flower scent — Participants in the experimental group will be informed about the effects of lavender scent on sleep and lavender sachets will be given. They will be informed that they should put these lavender sachets in their pillows every day and sleep with a lavender sachet for the next month, and that they should not make any changes in their rooms or beds other than the lavender sachet.
  Arms: Dry lavender flower scent

SUMMARY:
With aging, deterioration in sleep structure and balance occurs. In particular, individuals over the age of 65 often have sleep problems, and non-pharmacological methods used to solve this problem are much more reliable than pharmacological methods. It is important for nurses who contribute most to their care to regulate and facilitate sleep, which is one of the basic needs of people. Thanks to this study, it is planned to solve the sleep-related problems of elderly individuals by using the sedative and relaxing effect of the lavender plant, which is used in many areas, thus increasing their quality of life, and it is planned to prevent falls by increasing their physical balance controls. This study aims to determine the effect of lavender scent recommended for the elderly in Konya on sleep quality and physical balance. This research is a randomized experimental design with pretest-posttest control group. The research is planned to be carried out between January 2023 and November 2023. The population of the research consists of elderly individuals living in society. In order to determine the sample size, power

analysis will be made using the G-Power (v3.1.9.2) program. Personal Information Form and Pittsburgh Sleep Quality Index will be used in

data collection. The data obtained as a result of the research; It will be analyzed with IBM SPSS program. p<0.05 will be considered statistically

significant.

DETAILED DESCRIPTION:
The research data is planned to be collected between January 2023 and November 2023. Data will be collected from elderly individuals from the community. After the elderly individuals who meet the appropriate criteria are informed about the research, their verbal and written consent will be obtained that they agree to participate in the research.

Experimental Group In order to collect the pre-test data of the experimental group, individuals who accept the study will be asked to fill in the Personal Information Form, Sleep Quality Scale and Berg Balance Scale. The forms will be collected after the individuals mark the options closest to them on the forms. It is planned to last approximately 25-30 minutes. It is planned to recommend lavender scent as a nursing intervention to improve sleep quality in individuals with irregular sleep and low sleep quality. Participants in the experimental group will be informed about the effects of lavender scent on sleep and will be given lavender pouches. They will be informed that they should put these lavender pouches in their pillows where they sleep every day and that they should sleep with the lavender pouch for the next month, and that they should not make any changes in their rooms or beds other than the lavender pouch. After the one-month lavender scent application of the experimental group is completed, the post-test data will be collected for the experimental group. After the individuals who gave the closest answer to themselves completed the forms, the post-test data will be collected and the data collection phase of the research will be completed.

Control Group The study will start by collecting the pre-test data of the control group. Individuals who agree to participate in the study will be asked to fill in the Personal Information Form, Sleep Quality Scale and Berg Balance Scale to collect pre-test data. The forms will be collected after the individuals mark the options closest to them on the forms. After collecting the pre-test data, no intervention will be made to the participants for one month. At the end of one month, the control group will be administered the post-test with the same data collection tools.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the study.
* Working in shifts for at least three months
* Individuals who do not have a disease that would prevent research and communication will be included in the research.

Exclusion Criteria:

* Lavender allergy
* Patients with asthma, bronchitis
* Use of drug(s) that induce sleep
* Individuals who have received a medical diagnosis for attention will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-04-23 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Comparison of the effect of lavender scent on the experimental group according to the Pittsburgh Sleep Quality Index | At the end of 1 month
  The participants in the experimental group will be asked to put the lavender-scented sacs inside their pillows during sleep hours. Here, it is aimed to provide sleep order by taking advantage of the relaxing effect of the scent of lavender. After this application, the effect of lavender on sleep will be followed.
Determination of the effect of lavender odor on the balance control of the experimental group | At the end of 1 month
  The experimental group will be given a balance test before and after the lavender scent. The differences between the results will be tried to be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Berna Bayır, Principal Investigator — KTO Karatay University
Locations (1):
- Berna Bayır, Karatay, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No